CLINICAL TRIAL: NCT05058794
Title: Effects of Blood Flow Restriction Training vs Traditional Exercise in Patients With Knee Osteoarthritis.
Brief Title: Comparison Among the Effects of Blood Flow Restriction Training and Conventional Exercise in Knee Osteoarthritis.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REC/00947 Farah Anwar
Record Dates: First submitted 2021-09-17; First posted 2021-09-28 (Actual); Last update posted 2022-03-23 (Actual); Status verified 2022-03

CONDITIONS: Osteoarthritis, Knee; Hypertrophy
Keywords: Osteoarthritis; Blood Flow Restriction; Quadriceps; Resistance Training
MeSH Terms: conditions — Osteoarthritis, Knee; Hypertrophy; Osteoarthritis | interventions — Resistance Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Resistance exercise group (Experimental): During each exercise, only blood flow in the involved leg was restricted using an aneroid sphygmomanometer. Prior to exercise the cuff was placed on the most proximal portion of the limb and LOP was calculated in the body position that the blood flow restriction (BFR) stimulus would be applied. BFR pressure was set at 50% occlusion.Resistance applied for 1 minute (60 sec) with 30 % load of 1 repetition maximum. Subjects will receive treatment bilaterally.Participants will perform exercises 2 sets with 15 repetitions through 0 to 90 degrees.
  Secondly, Rest between sets (1 min) Therapist will help these positions to maintain Knee extension and Wall Squatting.
  The study includes interventional protocol of 6 weeks. Total sessions will be 12 and in each week there will 2 sessions with alternative days and follow up.
  Interventions: Other: Blood flow Restriction/Resistance Training
- Conventional Therapy Group (Active Comparator): Patients in this group will receive treatment via Knee extension,Wall squatting Each training session includes 3 minutes warm-up.First, participants will perform 2 sets with 15 repetitions in (0 to 90 degree.) Secondly, Rest between sets (1 min) Resistance applied for 1 minute (60 sec) with 30 % load of 1 repetition maximum. Subjects will receive treatment bilaterally. The study includes interventional protocol of 6 weeks. The sessions will be given on 2 alternate days making it a total of 12 sessions and then follow up.
  Interventions: Other: Conventional Therapy Group

INTERVENTIONS:
Other: Blood flow Restriction/Resistance Training — During each exercise, only blood flow in the involved leg was restricted using an aneroid sphygmomanometer. Prior to exercise the cuff was placed on the most proximal portion of the limb and limb occlusion pressure (LOP) was calculated in the body position that the Blood flow Restriction (BFR) stimulus would be applied. Blood Flow Restriction BFR pressure was set at 50% occlusion. Resistance applied for 1 minute (60 sec) with 30 % load of 1 repetition maximum. Subjects will receive treatment bilaterally. Participants will perform exercises 2 sets with 15 repetitions through 0 to 90 degrees.
  Arms: Resistance exercise group
Other: Conventional Therapy Group — Resistance applied for 1 minute (60 sec) with 30 % load of 1 repetition maximum. Subjects will receive treatment bilaterally.participants will perform 2 sets with 15 repetitions in (0 to 90 degree.)
  Arms: Conventional Therapy Group

SUMMARY:
The main objective of the study is to compare the effects of Blood flow Restriction training vs. traditional exercises on knee pain , knee functional disability and on quadriceps strength in patient with knee osteoarthritis.

DETAILED DESCRIPTION:
Osteoarthritis is a degenerative disease affecting the most commonly weight bearing joint.The common form of arthritis is osteoarthritis (OA) causing structural changes in the joint. Age is a common factor affecting the strength and muscle mass.Worldwide there is a drastic increase of osteoarthritis in the older population. In the past 20 years the prevalence of knee pain increased and reached up to 50% in the older population. The most common OA affecting lower extremity is in the knee Joint.Majority of the people affected by knee OA are the older population. Knee Joints being the most weight bearing joint affected in OA causing pain , limiting function and mobility.Mobility and function may be affected in osteoarthritic population usually experience pain and stiffness.

The main objective of this study is to compare the Effects of blood Flow restriction training vs conventional treatment exercises on knee pain, functional disability and quadriceps strengthening.

The main purpose of this study is to improve the muscular strength of lower limbs which are being affected in a disease osteoarthritis in the adult population.

ELIGIBILITY:
Inclusion Criteria:

* Pain : Subjects having unilateral or bilateral pain
* Pain type : subjects having chronic pain
* Includes diagnosed cases of knee osteoarthritis
* grades 2-3 according to the Kellgren and Lawrence method of grading
* Includes knee osteoarthritis patients with lateral tracking of patella which will assessed through Q angle test

Exclusion Criteria:

* Any other orthopaedic or neurological condition of hip and knee
* Sign and symptoms of lower motor neuron disease
* Current use of medication
* Radiculopathy
* Fracture
* Malignancy
* Thromboembolism
* Decreased range of motion

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2021-10-10 (Actual); Primary Completion 2022-02-11 (Actual); Study Completion 2022-02-11 (Actual)

PRIMARY OUTCOMES:
Muscle strength | 6 weeks
  Measurement of Quadriceps strength with portable weight machine.
Thigh Girth | 6 weeks
  Participants will be supine lying and knee in extension, standing or knee at 90 degree. Proximal to the patellar pole superiorly one measurement with a non-elastic tape at the inguinal fold, then mark the mid-point at the mid-thigh level measuring in centimeters/inches.
Numeric Pain Rating Scale ( NPRS) | 6 weeks
  Patient will be asked if there is any pain in knee from the scale of 0 to 10.
Q angle Measurement | 6 weeks
  Subject will be in supine position with knee extension and quadriceps are relaxed, examiner will measure the q angle with flexible inch tape and goniometer. The Q- angle is measured by extending a line through the center of the patella to the anterior superior iliac spine and another line from the tibial tubercle through the center of the patella.

CONTACTS AND LOCATIONS:
Overall Officials: Saad Rauf, Master, Principal Investigator — Riphah International University
Locations (2):
- Pakistan (2):
  - Gulberg Medical Complex, Islamabad, Federal
  - Medcity International Hospital, Islamabad, Federal

IPD SHARING:
Plan to Share IPD: No